CLINICAL TRIAL: NCT06818708
Title: A Randomized, Single-Blinded, Sham-Controlled Study Evaluating the Efficacy and Safety of RELAY, a Device Enabling Both Local Anesthetic Delivery and Neuromodulation Following Shoulder or Foot Surgery: Single Arm Training Run-In Phase
Brief Title: Feasibility of an Analgesic Device Enabling Local Anesthetic Delivery and Neuromodulation After Shoulder/Foot Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Gate Science (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RELAY Feasibility
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Rotator Cuff Injuries; Shoulder Disease; Hallux Valgus; Ankle Arthropathy
MeSH Terms: conditions — Rotator Cuff Injuries; Hallux Valgus

STUDY DESIGN:
Intervention Model Description: A series of participants all receiving active treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental Treatment (Experimental): RELAY catheter will be inserted under ultrasound guidance followed by a local anesthetic bolus injection. If a patient's surgeon requests a postoperative continuous peripheral nerve block, a ropivacaine 0.2% infusion will be initiated in the recovery room. Within the recovery room, the stimulators will be connected to participants' phones and turned on. The catheters will be removed on postoperative day 7.
  Interventions: Device: Experimental Treatment

INTERVENTIONS:
Device: Experimental Treatment — Percutaneous peripheral nerve stimulation with a frequency between 1-250 Hz, a pulse duration of 1-200 µs, and a current of 0.001-10 mA (1-10,000 µA). If the same pattern holds for the RELAY device as for previously tested peripheral nerve stimulators, we will maximize frequency, minimize pulse duration, and have participants adjust the amplitude, as needed.
  Other Names: percutaneous peripheral nerve stimulation

SUMMARY:
Postoperative pain remains undertreated with inadequate analgesic options. Opioids have well-known limitations for both individuals and society; single-injection and continuous peripheral nerve blocks provide intense analgesia but are limited in duration to 24-72 hours; and current neuromodulation options-with a duration measured in weeks and not hours-are prohibitively expensive and require an additional procedure. One possible solution is a device currently under investigation to treat postoperative pain. The RELAY system (Gate Science, Moultonborough, New Hampshire) is comprised of a basic catheter-over-needle device to allow administration of a single-injection of local anesthetic via the needle (or catheter) followed by a perineural local anesthetic infusion via the remaining catheter (when desired). Subsequent to the local anesthetic administration, instead of removing the catheter as with all previous continuous peripheral nerve block equipment, electric current may be delivered via the same catheter and an integrated pulse generator for up to 28 days. This is potentially revolutionary because it would allow an anesthesiologist to deliver (1) a single-injection peripheral nerve block; (2) a continuous peripheral nerve block; and (3) neuromodulation using a single device that can theoretically be placed in the same amount of time required for a single-injection peripheral nerve block. Instead of providing fewer than 24 hours of postoperative analgesia, up to 28 days of pain control could be delivered without disruption of existing practice patterns. The ultimate objective of the proposed investigation is to prepare for a randomized clinical trial investigating the use of the RELAY device to provide postoperative analgesia.

This feasibility study will be a series of participants all receiving both local anesthetic and electric current via a single device (RELAY, Gate Science, Moultonborough, New Hampshire). The purpose will be to optimize the insertion approach and stimulation administration during the first 7 days following foot and shoulder surgery as well as training the clinical investigators.

DETAILED DESCRIPTION:
Specific Aim: To determine the feasibility and optimize the protocol for the RELAY device following foot and shoulder surgery to prepare for the subsequent randomized, controlled pilot study.

For individuals of childbearing potential, a sample of urine will be collected before any study interventions to confirm a non-pregnant state (this is standard procedure for all surgical patients). The RELAY device combines a catheter-over-needle to permit ultrasound-guided percutaneous insertion with the tip adjacent to a peripheral nerve or plexus, followed by needle removal which leaves the catheter in situ to deliver a bolus of local anesthetic (if desired) and subsequent perineural local anesthetic infusion (if desired). The catheter also has 3 integrated electrodes to enable neuromodulation using the integrated pulse generator and battery.

Participants will have standard external monitors placed and oxygen delivered by facemask or nasal cannula. The peripheral nerve block site(s) will be cleansed with chlorhexidine gluconate and isopropyl alcohol. Intravenous sedation/analgesia with midazolam and/or fentanyl will be titrated for patient comfort as is standard for peripheral nerve block administration. The nerves treated will include the sciatic proximal to the popliteal crease for foot surgery and the brachial plexus for shoulder surgery. The target nerve(s) will be visualized with ultrasound using a transverse cross-sectional (short axis) view and a skin wheal of local anesthetic will be raised inferior to the transducer to anesthetize the skin and then the track towards the target. The RELAY with the integrated needle will be inserted adjacent to the target nerve with an in-plane approach. Dextrose 5% in water (1-20 mL) will be injected via the needle to open a space around the target nerve(s), the catheter advanced, and the needle subsequently withdrawn.

Electrical current will be introduced with increasing intensity via each of the anode electrodes to optimize participant's perceived stimulation (control provided by the Gate Keeper app from an investigator's phone or tablet). Accurate lead placement will be confirmed with subject reports of comfortable sensations over the surgical site without eliciting muscle contractions. The minimum threshold and maximum comfortable amplitudes will be determined along with the optimal frequency, pulse duration, and anode/cathode. Starting from the lowest possible current the investigators increase the current until the participant states that they feel a "buzzing" sensation (some describe it as a "comfortable massage"). That is the minimal sensed current. The investigators then continue increasing with the instructions to let us know when it starts to be less comfortable-and to stop us before it hurts. That is the maximum comfortable current. The stimulator will be then set to deliver the minimum threshold amplitude and turned off for surgery. The pulse generator of the RELAY has a frequency between 1-250 Hz, a pulse duration of 1-200 µs, and a current of 0.001-10 mA (1-10,000 µA). The investigators will maximize frequency, minimize pulse duration, and have participants adjust the amplitude following surgery, as needed.

Local anesthetic (10 mL of lidocaine 2% with epinephrine) will be injected with negative aspiration every 3 mL and resulting sensory block confirmed to ensure accurate catheter tip placement. Following block confirmation (sensory deficits in the expected nerve distributions), the RELAY will be affixed with both surgical adhesive (2-Octyl 2-cyanoacrylate) at the entry site and a chlorohexidine-impregnated occlusive dressing [research specific]. Subsequently, 10 mL of bupivacaine 0.5% with epinephrine will be injected negative aspiration every 3 mL along with a supplemental single-injection saphenous nerve block for foot/ankle surgery.

Intraoperatively, surgeons will be permitted to infiltrate the surgical area with long-acting local anesthetic as their common practice dictates.

Postoperatively, the stimulators will be connected to participants' phones and turned on. If a patient's surgeon requests a postoperative continuous peripheral nerve block, a ropivacaine 0.2% infusion will be provided per standard UC San Diego protocol. After 7 days, participants themselves or their caretaker will remove the occlusive dressing and withdraw the catheter (and integrated electrodes) with gentle traction and rotation at home. The devices are single-use and disposable.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants of at least 18 years of age
2. Undergoing a rotator cuff repair, total shoulder arthroplasty, ankle arthroplasty/arthrodesis, or foot surgery anticipated to result in moderate-to-severe pain for at least one week
3. Planned single-injection peripheral nerve block(s)
4. An Android or Apple smartphone able to download the Gate Keeper controller app

Exclusion Criteria:

1. Chronic opioid or tramadol use (daily within prior 2 weeks and duration > 4 weeks)
2. Neuro-muscular deficit of the surgical limb
3. Compromised immune system based on medical history (e.g., immunosuppressive therapies such as chemotherapy, radiation, sepsis, infection), or other conditions that places the subject at increased risk of infection
4. Implanted spinal cord stimulator, cardiac pacemaker/defibrillator, deep brain stimulator, or other implantable neurostimulator whose stimulus current pathway may overlap
5. History of bleeding disorder
6. Antiplatelet or anticoagulation therapies other than aspirin
7. Allergy to skin-contact materials (occlusive dressings, bandages, tape etc.)
8. Incarceration
9. Pregnancy
10. Moderate pain (NRS > 3) in an anatomic location other than the surgical site
11. Anxiety disorder
12. History of substance misuse
13. Inability to communicate with the investigators
14. Inability to contact the investigators during the treatment period, and vice versa (e.g., lack of telephone access)
15. Allergy to amide local anesthetics
16. Morbid obesity (body mass index > 40 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, Ms, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ilfeld BM, Said ET, Park BH, Sinha SK, Leek B, Meunier MJ, Foran IM, Hurvitz A, Kent WT, Schwartz AK, Abdullah B, Alkabalan R, Lau N, Finneran JJ. Percutaneous analgesic device enabling both local anesthetic delivery and electrical stimulation (neuromodulation) of peripheral nerves: a pilot feasibility study (case series). Reg Anesth Pain Med. 2025 Sep 25:rapm-2025-107029. doi: 10.1136/rapm-2025-107029. Online ahead of print. PMID 41005804
- See also: article containing the results — https://rapm.bmj.com/content/rapm/early/2025/09/25/rapm-2025-107029.full.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Treatment
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20
Height [Mean (Standard Deviation); unit: cm] | 173 (9)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 87 (20)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30 (6)

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Pain Intensity 1st Week
Description: The median of 5 daily "average" pain intensity scores for Days 1-4 and 7 as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Time Frame: Days 1-4 and 7
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
units on a scale | 2 [0 to 3]

2. Secondary Outcome: Cumulative Opioid Use 1st Week
Description: The cumulative opioid use measured in oxycodone equivalents during the first 7 days following surgery
Time Frame: The first 7 days following surgery
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
milligrams | 43 [18 to 73]

3. Secondary Outcome: Brief Pain Inventory (Interference Sub Scale) Day 3
Description: The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale; (2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include solely the interference subscale with a minimum score of 0 (optimal outcome) and maximum score of 70 (worst possible outcome).
Time Frame: Postoperative day 3
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
units on a scale | 2 [0 to 4]

4. Secondary Outcome: Brief Pain Inventory (Interference Sub Scale) Day 7
Description: as for outcome 3
Time Frame: Postoperative day 7
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
units on a scale | 0 [0 to 7]

5. Secondary Outcome: Worst Daily Pain Intensity 1st Week
Description: The median of 5 daily "worst" (maximum) pain intensity scores for Days 1-4 and 7 as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Time Frame: Days 1-4 and 7
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
units on a scale | 4.0 [2.6 to 6.0]

6. Secondary Outcome: Awakenings Due to Pain 1st Week
Description: Cumulative number of nightly awakenings due to pain
Time Frame: Collected on postoperative days 1, 2, 3, 4, and 7
Measure: Median (Inter-Quartile Range); unit: number of awakenings
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
number of awakenings | 2 [0 to 7]

7. Secondary Outcome: Average Daily Pain Intensity Day 7
Description: The "average" pain intensity score on Day 7 as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Time Frame: Day 7
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
units on a scale | 0 [0 to 1.1]

8. Secondary Outcome: Worst (Maximum) Daily Pain Intensity Day 7
Description: The "worst" pain intensity score on Day 7 as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Time Frame: Day 7
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
units on a scale | 1.8 [1.0 to 3.5]

9. Secondary Outcome: Opioid Consumption Day 7
Description: The cumulative opioid use from the previous 24 hours measured in oxycodone equivalents as recorded on Day 7
Time Frame: Day 7
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
milligrams | 0 [0 to 0]

10. Secondary Outcome: Daily "Average" Pain Intensity
Description: The "average" pain intensity score on each postoperative day as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Time Frame: postoperative Days 1, 2, 3, 4, 7, 8 and 14
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
units on a scale
  Day 1 | 3 [1 to 4.3]
  Day 2 | 2 [.9 to 3.3]
  Day 3 | 2 [0 to 3]
  Day 4 | 1 [0 to 2.3]
  Day 7 | 0 [0 to 1.1]
  Day 8 | 0 [0 to 1.1]
  Day 14 | 0 [0 to 1.3]

11. Secondary Outcome: Daily "Worst" Pain Intensity
Description: The "worst" pain intensity score on each postoperative day as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Time Frame: postoperative Days 1, 2, 3, 4, 7, 8 and 14
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
units on a scale
  Day 1 | 5 [4 to 7.1]
  Day 2 | 4.5 [3.1 to 6.3]
  Day 3 | 4.3 [3.3 to 6]
  Day 4 | 3 [.4 to 4]
  Day 7 | 1.8 [1 to 3.5]
  Day 8 | 2 [0 to 3]
  Day 14 | 2 [0 to 4]

12. Secondary Outcome: Daily Opioid Consumption
Description: The cumulative opioid use from the previous 24 hours measured in oxycodone equivalents as recorded on Days 1-4, 7, 8, and 14
Time Frame: postoperative Days 1, 2, 3, 4, 7, 8 and 14
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 20
milligrams
  Day 1 | 0.3 [0 to 2]
  Day 2 | 0 [0 to 1.3]
  Day 3 | 0 [0 to 1]
  Day 4 | 0 [0 to 0]
  Day 7 | 0 [0 to 0]
  Day 8 | 0 [0 to 0]
  Day 14 | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Experimental Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Treatment (N=20)
Baton separation from pulse generator during intentional removal (Surgical and medical procedures) | 1 (1)
Perineural catheter occlusion (Surgical and medical procedures) | 3 (3)
Accidental catheter dislodgment (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT06818708/Prot_SAP_000.pdf